CLINICAL TRIAL: NCT02313441
Title: Cardio- and Reno-protective Effect of Remote Ischemic Preconditioning in Patients Undergoing Percutaneous Coronary Intervention. A Prospective, Non-randomized Controlled Trial.
Brief Title: Cardio- and Renoprotective Effect of Remote Ischemic Preconditioning in Patients Undergoing Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Khairy Mohamed Hassan, Dr., Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIPC1
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease
Keywords: remote ischemic preconditioning
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC (Remote Ischemic Pre-Conditioning) (Active Comparator): Patients used RIPC had a blood pressure cuff placed around their upper arm at < 2 hours before the PCI procedure. The blood pressure cuff was inflated to for 5 minutes, followed by 5 minutes of deflation. This procedure was repeated 3 times
  Interventions: Other: Remote Ischemic Pre-Conditioning
- Control (Placebo Comparator): Control participants did not experience this procedure of transient upper-limb ischemia.
  Interventions: Other: Remote Ischemic Pre-Conditioning

INTERVENTIONS:
Other: Remote Ischemic Pre-Conditioning — The blood pressure cuff was inflated to a pressure of 200 mm Hg for 5 minutes, followed by 5 minutes of deflation to allow reperfusion. This procedure was repeated 3 times by the resident doctors in the pre-cath room

SUMMARY:
Myocyte necrosis occurs frequently in elective percutanious percutaneous coronary intervention (PCI) and is associated with subsequent cardiovascular events. This study assessed the cardio- and reno-protective effect of remote ischemic preconditioning (RIPC) in patients undergoing elective PCI. 200 patients were randomized into 2 groups: 100 patients received RIPC (created by three 5-minute inflations of a blood pressure cuff to 200 mm Hg around the upper arm, separated by 5-minute intervals of reperfusion) < 2 hours before the PCI procedure, and the control group (n = 100).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 85 years of age,
* scheduled to undergo an elective PCI and
* able to give an informed consent were eligible for enrollment in the study.
* Elective PCI was defined as any coronary revascularization in a low-risk patient who presents to the facility for a planned PCI or for a coronary angiogram followed by ad hoc PCI.

Exclusion Criteria:

* (1) emergency PCI, (2) baseline troponin value ≥ 0.04 ng/mL, (3) nicorandil or glibenclamide use (preconditioning-mimetic and preconditioning-blocking medication, respectively), (4) those who could not give informed consent, and (5) patients with severe renal impairment or on regular dialysis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of PCI- related myocardial infarction (MI 4a) at 24 hours after PCI. | 24 hours
  PCI-related myocardial infarction (MI 4a) was defined as cardiac Troponin I (cTnI) elevation >0.20ng/mL (5 times the upper reference limit) 24 hr. post PCI.

SECONDARY OUTCOMES:
incidence of contrast induced nephropathy (CIN) at 72 hours after contrast exposure | 72 hours
  CIN was defined as an increase in the serum creatinine level of more than 0.5 mg/dl or more than 25 % from baseline within 3 days after procedure without any other identifiable cause of acute kidney injury.

OTHER OUTCOMES:
Chest pain severity during PCI | 1 hours
  Chest pain severity during PCI was graded on a scale of 0 for no pain to 10 for the most severe discomfort ever experienced
level of C-reactive protein (CRP)24 hr post PCI | 24h post procedure
  C-reactive protein level was measured 24 hr. post PCI to assess the inflammatory response .
major adverse events (MAE) at 3 month follow up | 90 days Follow-up
  Death was defined as "all-cause" death at follow-up. Acute coronary syndrome (ACS) was defined using standard diagnostic criteria. Heart failure (HF) during follow-up, was defined as either the presence of rales in more than one third of the lung fields that did not clear with coughing or evidence of pulmonary oedema on chest radiograph. Hemodialysis as a complication of acute deterioration of renal function post PCI was also calculated. Only the most serious event of MAE was used to calculate the cumulative MAE per patient according to the following sequence: death>ACS > HF> Hemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman KM Hassan, MD. PhD., Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

REFERENCES:
- [Background] Ali ZA, Callaghan CJ, Lim E, Ali AA, Nouraei SA, Akthar AM, Boyle JR, Varty K, Kharbanda RK, Dutka DP, Gaunt ME. Remote ischemic preconditioning reduces myocardial and renal injury after elective abdominal aortic aneurysm repair: a randomized controlled trial. Circulation. 2007 Sep 11;116(11 Suppl):I98-105. doi: 10.1161/circulationaha.106.679167. PMID 17846333
- [Background] Hoole SP, Heck PM, Sharples L, Khan SN, Duehmke R, Densem CG, Clarke SC, Shapiro LM, Schofield PM, O'Sullivan M, Dutka DP. Cardiac Remote Ischemic Preconditioning in Coronary Stenting (CRISP Stent) Study: a prospective, randomized control trial. Circulation. 2009 Feb 17;119(6):820-7. doi: 10.1161/CIRCULATIONAHA.108.809723. Epub 2009 Feb 2. PMID 19188504